CLINICAL TRIAL: NCT03143608
Title: Laparoscopic Hiatal Hernia Repair Followed Immediately By Transoral Incisionless Fundoplication Using the Esophyx Device: Efficacy And Safety In 99 Patients In A Community Setting
Brief Title: GERD Treatment With Transoral Incisionless Fundoplication (TIF) Following Hiatal Hernia Surgery
Acronym: GERD
Status: Completed | Type: Observational
Sponsor: Peter G Mavrelis (Individual)
Responsible Party: Sponsor-Investigator, Peter G Mavrelis, Gastroenterologist, Mavrelis, Peter G., M.D.
Organization: Mavrelis, Peter G., M.D. (Individual)
Other Study IDs: 04/03/2014
Record Dates: First submitted 2017-04-29; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Gastro Esophageal Reflux
Keywords: GERD; Hiatal hernia repair; Transoral Incision less fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Indiana group: 50 adult patients males and females with GERD and 2-5 cm hiatal hernias. Each had laparoscopic hiatal hernia repair followed by transoral incisionless fundoplication
  Interventions: Device: Esophyx
- Wisconsin group: 49 adult patients males and females with GERD and 2-5 cm hiatal hernias. Each had laparoscopic hiatal hernia repair followed by transoral incisionless fundoplication
  Interventions: Device: Esophyx

INTERVENTIONS:
Device: Esophyx — Laparoscopic hiatal hernia repair followed immediately by transoral incisionless fundoplication under general anesthesia using the Esophyx device

SUMMARY:
The investigators prospectively studied ninety nine GERD patients following laparoscopic hiatal surgery combined with transoral incisionless fundoplication at two community hospitals. General surgeons and gastroenterologists participated in the study. GERD questions were recorded before and at six and twelve months.

DETAILED DESCRIPTION:
GERD unresponsive to medical therapies can be treated by laparoscopic Nissen fundoplication or endoluminal techniques. The investigators have extensive experience with Transoral Incisionless Fundoplication(TIF). TIF is not indicated in patients with a hiatal hernia larger than 2 cm. Performing a Hiatal Hernia Repair(HHR) in those cases will make a patient eligible for TIF. HHR followed immediately by the TIF procedure under the same anesthetic session is called a Hybrid-TIF (HTIF). The study examines the safety and efficacy of this approach.

Prospective data were collected from patients who underwent HTIF at two 300 bed community hospitals. Questionnaires were administered before the procedure, and mailed at 6 and 12 mos. They were the GERD-HRQL-health related quality of life, RSI-reflux symptom index, and GSRS-gastrointestinal symptom rating scale.

The study continues with the new Esophyx-Z device

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical or atypical GERD who want a surgical solution to control symptoms.
* Patients need a 2-5 cm hiatal hernia and have a BMI of less than 36.

Exclusion Criteria:

* Hiatal hernias larger than 5 cm and BMI greater than 36.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with GERD
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Control of GERD symptoms | one year
  GERD health related quality of life questionnaire
Control of GERD symptoms | one year
  Reflux symptom index questionnaire
Control of GERD symptoms | one year
  Gastrointestinal symptom rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mavrelis, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Methodist Hospital, Merrillville, Indiana
  - Affinity Health System, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
presentation at national meeting

REFERENCES:
- [Result] Ihde GM, Besancon K, Deljkich E. Short-term safety and symptomatic outcomes of transoral incisionless fundoplication with or without hiatal hernia repair in patients with chronic gastroesophageal reflux disease. Am J Surg. 2011 Dec;202(6):740-6; discussion 746-7. doi: 10.1016/j.amjsurg.2011.06.035. Epub 2011 Oct 20. PMID 22014853